CLINICAL TRIAL: NCT05139940
Title: Validation of Artificial Intelligence Enabled TB Screening and Diagnosis in Zambia
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Other Study IDs: Google AI
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
Keywords: Screening; Diagnosis; Artificial Intelligence; Chest X-ray
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pilot Group to calibrate the operating points for AI algorithms (Estimated Enrollment up to 500): Diagnostic Test: TB AI algorithm performance in detecting active TB.
  Diagnostic Test: TB diagnosis from sputum and urine (Smear microscopy, Xpert MTB RIF/ultra, Lipoarabinomannan (LAM) and mycobacterial culture)
  Diagnostic Test: Abnormal/Normal AI algorithm to detect abnormal/normal CXRs.
  Diagnostic Test: Radiologist evaluation of CXRs for active TB, abnormal/normal.
  Diagnostic Test: Labs: Hemoglobin level, HIV status, CD4 count.
- Main Cross Sectional Group (Estimated Enrollment 1932 minus the volume in pilot): Diagnostic Test: TB AI algorithm performance in detecting active TB.
  Diagnostic Test: TB diagnosis from sputum and urine (Smear microscopy, Xpert MTB RIF/ultra, Lipoarabinomannan (LAM) and mycobacterial culture)
  Diagnostic Test: Abnormal/Normal AI algorithm to detect abnormal/normal CXRs.
  Diagnostic Test: Radiologist evaluation of CXRs for active TB, abnormal/normal.
  Diagnostic Test: Labs: Hemoglobin level, HIV status, CD4 count.

SUMMARY:
Tuberculosis (TB) is a global epidemic and for many years has remained a major cause of death throughout the developing world. Zambia is among the top 30 TB/HIV high burden countries. Chest X-ray (CXR) is recommended as a triaging test for TB, and a diagnostic aid when available. However, many high-burden settings lack access to experienced radiologists capable of interpreting these images, resulting in mixed sensitivity, poor specificity, and large inter-observer variation. In recognition of this challenge, the World Health Organization has recommended the use of automated systems that utilize artificial intelligence (AI) to read CXRs for screening and triaging for TB. In this study, we primarily evaluate the performance of our AI algorithm for TB, and secondarily for Abnormal/Normal.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 18 years and older with a known HIV status or are willing to undergo HIV testing if unknown HIV status and meet the following criteria will be included in the study:

  * Presumptive TB patients defined as having any of the following:

    ○ Cough, Weight loss, Night sweats, Fever
  * Household /close TB contacts regardless of symptoms
  * Newly diagnosed HIV regardless of symptoms.

Exclusion Criteria:

* Individuals who do meet the above inclusion criteria will be excluded. In addition, individuals with history of TB treatment within 365 days prior to enrolment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted from Chainda South Clinic, Chawama and Kanyama General Hospitals. These facilities are selected based on existing access to digital radiography. Participants will be drawn from patients attending these health facilities for:
  * Health services
  * TB households of those who are close contacts of TB households within the catchment area of these facilities
Sampling Method: Non-Probability Sample
Enrollment: 2432 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Pilot Group to calibrate the operating points for AI algorithms | 2 months
  1. Operating point selection for TB AI algorithm and Abnormal/Normal AI algorithm on CXRs for outcomes listed in Main Cross Sectional Group.
Main Cross Sectional Group | 7 months
  1. TB AI algorithm sensitivity and specificity in detecting active TB on CXR compared to panel of radiologists

SECONDARY OUTCOMES:
Main Cross Sectional Group: | 7 months
  1. TB AI algorithm sensitivity and specificity in detecting active TB compared to World Health Organisation (WHO) performance guidelines of 90% sensitivity and 70% specificity
Main Cross Sectional Group | 7 months
  2. Abnormal/Normal AI algorithm sensitivity and specificity compared to 90% sensitivity and 50% specificity.

CONTACTS AND LOCATIONS:
Locations (3):
- Zambia (3):
  - Chainda South Health Facility, Lusaka, Lusaka Province
  - Chawama first level hospital, Lusaka, Lusaka Province
  - Kanyama level 1, Lusaka, Lusaka Province